CLINICAL TRIAL: NCT04663737
Title: A Phase II, Randomized and Controlled Investigator Initiated Trial Evaluating Safety, Pharmacokinetics and Clinical Benefit of Silmitasertib (CX-4945) in Outpatient Adult Subjects With Moderate Coronavirus Disease 2019 (COVID-19)
Brief Title: Evaluating Safety, Pharmacokinetics and Clinical Benefit of Silmitasertib (CX-4945) in Subjects With Moderate COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Senhwa Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CX4945 AV01-IIT
Record Dates: First submitted 2020-12-01; First posted 2020-12-11 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: Covid19
Keywords: Moderate Covid19
MeSH Terms: conditions — COVID-19 | interventions — silmitasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A will receive the best supportive care and/or recommended standard of care (at this point no standard of care drugs are recommended by CDC for patients with moderate COVID-19) in combination with the study drug Silmitasertib
  Interventions: Drug: Silmitasertib
- Group B (Active Comparator): Group B (control) that will receive the same care as the Group A but without Silmitasertib
  Interventions: Drug: SOC

INTERVENTIONS:
Drug: Silmitasertib — Capsules
  Other Names: CX-4945
  Arms: Group A
Drug: SOC — Some therapeutics for COVID-19 are available through EUA. SOC treatment availability is expected to change during the course of this trial.
  Other Names: SOC/ Best Supportive Care
  Arms: Group B

SUMMARY:
This single-center, open-label, 2 arm parallel-group, randomized, interventional prospective exploratory study in 20 subjects aimed to evaluate safety and explore putative clinical benefits of Silmitasertib 1000 mg BID dose in patients with moderate COVID-19. Two-arm trial comparing the SOC/supportive care alone to the SOC/supportive care with addition of Silmitasertib (allocation ratio 1:1).

DETAILED DESCRIPTION:
Silmitasertib is a first-in-class small molecule drug that targets Casein Kinase 2 (CK2). Protein kinase CK2 phosphorylates key proteins required to trigger mechanisms vital for viral replication and also is involved in development of host anti-viral immune response. SARS-CoV-2 viral proteins interacting with many human host proteins affect multiple innate immune pathways. One of these key proteins dysregulated by SARS-CoV-2 is the protein kinase CK2. SARS-COV-2 upregulates CK2 to support viral replication, avoid innate immune response and spread virus to nearby cells. Overactivation of CK2 indirectly contribute to successful viral replication and development of cytokine storm.SARs-Cov-2-induced overexpression of CK2, while pharmacological inhibition of CK2 suppresses virus proliferation. CK2 signaling appears to be an important pathway hijacked by SARS-CoV-2.

Emerging pre-clinical and clinical data and results of independent efficacy evaluation conducted by Utah State University and UCSF COVID-19 research group and Senhwa Biosciences hypothesize that Silmitasertib (CX-4945) could potentially quell virus-provoked aberrant hyperactivation of the innate immune system by inhibition of upregulated CK2 protein kinase, preferentially restoring normal host cell cytokine regulation, and attenuating viral replication in patients with moderate to severe COVID-19, thereby preventing disease progression and improving clinical outcomes. Intended target patient population for treatment with Silmitasertib (CX-4945) are SARS-COV-2 positive patients with moderate to severe COVID-19, since in the moderate to severe stage of the disease infected cells actively produce viral proteins that dysregulate signaling pathways to allow viruses to manipulate host immune responses to create an environment more favorable for infection, that may not be observed in the initial or mild stage of the disease.

CX-4945 demonstrated remarkable clinical benefits under emergency IND authorization in a patient with COVID-19 pneumonia not responsive to remdesivir, dexamethasone and antibiotics and requiring supplemental oxygen. The patient recovered and was discharged from the hospital in five days of treatment with CX-4945.

The purpose of this open-label, randomized, 2 arm parallel-group controlled, interventional prospective exploratory study in 20 subjects is to evaluate safety, tolerability and pharmacokinetics of Silmitasertib (CX-4945) 1000 mg BID dose, to compare time to clinical recovery, and putative clinical benefit across treatment groups, and to evaluate anti-viral activities in COVID-19 patients.

Silmitasertib is a generally well-tolerated medication. Most adverse events reported were mild to moderate in severity. The most common toxicities associated with CX-4945 were gastrointestinal disorders, manageable with drug discontinuation or use of anti-diarrheal medication. Based on the currently available data, the identified or potential risks of the product do not outweigh its identified or potential benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female adult ≥ 18 years of age
2. Diagnosed with COVID-19 by standard RT-PCR assay or equivalent testing
3. Outpatient subjects with moderate illness caused by SARS-CoV-2 infection as defined below,

   * Symptoms of moderate systemic illness/infection with COVID-19:

   At least two of the key COVID-19-related symptoms with score 2 or higher (0=none, 1=mild, 2=moderate, and 3=severe): cough, sore throat, malaise, headache, muscle pain, fever, neurological symptoms such as brain fog/concentration challenges, gastrointestinal symptoms or shortness of breath with exertion

   AND
   * Clinical signs indicative of moderate systemic illness/infection with COVID-19 At least 1 of the following: respiratory rate ≥ 20 breaths per minute, heart rate ≥ 90 beats per minute

   AND
   * No clinical signs indicative of Severe or Critical Illness Severity required hospitalization (see exclusion criterion #1)
4. Patient (or legally authorized representative) provides written informed consent prior to initiation of any study procedures.
5. Adequate hematopoietic capacity, as defined by the following:

   1. Hemoglobin ≥ 9.0 g/dL and not transfusion dependent
   2. Platelets ≥ 100,000/mm3
   3. Absolute neutrophil count ≥ 1500 cells/mm3
6. Adequate hepatic function, as defined by the following:

   1. AST and ALT ≤ 2.5 times upper limit of normal (ULN)
   2. Total bilirubin ≤ 1.5 x ULN
   3. Albumin ≥ 3.0 g/dL
7. Adequate renal function, as defined by the following:

   a. Renal: calculated creatinine clearance >45 mL/min for patients with abnormal, increased creatinine levels (Cockcroft-Gault formula).
8. Ability to take oral medication and be willing to adhere to drug administration and premedication requirements (see Section 6.3) throughout study duration.

Exclusion Criteria:

1. Any signs indicative of Severe or Critical Illness Severity required hospitalization as defined below:

   * Severe COVID-19: Shortness of breath in rest, or respiratory distress, respiratory rate (RR) >/= 30 per minute, heart rate (HR) >/=125 bpm, SpO2</=93% on room air at sea level or PaO2/FiO2<300
   * Critical COVID-19: respiratory failure required mechanical ventilation, oxygen delivered by high-flow nasal cannula, ESMO; shock or multi-organ dysfunction/failure
2. Pregnant or nursing women. (NOTE: Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation. Should a man father a child, or a woman become pregnant or suspect she is pregnant while participating in this study, he or she should inform the treating physician immediately.)
3. Active or uncontrolled infections other than COVID-19 or with serious illnesses or medical conditions which would not permit the patient to receive study treatment
4. Chronic diarrhea (excess of 2-3 stools/day above normal frequency)
5. Concomitant treatment with another investigational drug from Day 1 through Day 28.
6. Current use or anticipated need for drugs that are known strong inhibitors or inducers of major CYP enzymes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris P. Recknor, MD, Principal Investigator — Center for Advanced Research and Education
Locations (1):
- Center for Advanced Research and Education, Gainesville, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 Nov 2020 - First Patient First Visit; 04 Oct 2021 - Last Patient Last Visit.
Groups:
- Group A: Group A will receive the best supportive care and/or recommended standard of care (at this point no standard of care drugs are recommended by CDC for patients with moderate COVID-19) in combination with the study drug Silmitasertib.
  Silmitasertib: Capsules 1000mg/BID
Period: Overall Study
Arm/Group | Group A | Group B
Started | 10 | 10
Completed | 8 | 10
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: The ITT population was defined as all randomized subjects. This population was used as the primary analysis population for analysis of the primary and secondary efficacy endpoints.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (14.18) | 50.7 (14.86) | 47.3 (14.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 7 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Study Site [Count of Participants; unit: Participants]
  001-CARE (Center for Advanced Research & Education) | 6 | 4 | 10
  002-CAR (CA's Research) | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) Within the CX-4945 Treatment Group
Description: To assess adverse events associated with the administration of CX-4945 orally, twice daily to patients with moderate COVID-19. The occurrence of overall AEs in the two treatment groups are summarized.
Time Frame: From randomization (Day 1) to Day 60
Population: Population: Safety Population; The Safety population is defined as any subject receiving at least one dose of CX-4945 or standard of care treatment after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
Participants | 9 | 4

2. Secondary Outcome: Clinical Recovery Associated With COVID-19 Within the CX-4945 Treatment Group
Description: To compare the number of days to clinical recovery specifically associated with COVID-19 in the CX-4945 treatment group as compared to the control arm by Day 14 of the study.
Time Frame: First 14 days of the study.
Population: 2 patients in Group A, 3 patients in Group B were censored from this analysis per protocol.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 7
Days | 7 [4 to 12] | 14 [7 to 14]

3. Secondary Outcome: Anti-Viral Activity of CX-4945
Description: To evaluate preliminary evidence of anti-viral activity of CX-4945 as compared to the control arm.
Time Frame: Quantitative changes in viral load from Day 1 to Day 28.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
Participants
  Viral Clearance Day 8: Negative | 4 | 6
  Viral Clearance Day 8: Positive | 3 | 2
  Viral Clearance Day 8: Inconclusive | 2 | 0
  Viral Clearance Day 8: Not Evaluated | 1 | 2
  Viral Clearance Day 14 (EOT): Negative | 5 | 7
  Viral Clearance Day 14 (EOT): Positive | 0 | 1
  Viral Clearance Day 14 (EOT): Inconclusive | 2 | 1
  Viral Clearance Day 14 (EOT): Not Evaluated | 3 | 1

4. Secondary Outcome: Maximum Plasma Concentration [Cmax] of CX-4945
Description: To evaluate the maximum plasma concentration of CX-4945 when given at 1000 mg BID PO (Experimental Arm taking CX-4945 only i.e. Group A).
Time Frame: Plasma sample of CX-4945 are collected at the following timepoints: Day 1: pre-dose, 1, 2, 3, 6 and 24 hours post Day 1 morning dose and Day 14: pre-dose, 1, 2, 3, 6, 24, 48 and 72 hours post Day 14 morning dose.
Population: Plasma sample of CX-4945 are collected from the first four subjects randomized to treatment arm A.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group A
Number analyzed (Participants) | 4
ng/mL
  Day 1 | 19035.99 (15918.33)
  Day 14: number analyzed (Participants) | 3
  Day 14 | 38749.51 (32469.52)

5. Secondary Outcome: Time to Maximum Observed Plasma Concentration [Tmax] of CX-4945
Description: To evaluate the time to maximum observed plasma concentration of CX-4945 when given at 1000 mg BID PO (Experimental Arm taking CX-4945 only i.e. Group A).
Time Frame: as for outcome 4
Population: Plasma sample of CX-4945 are collected from the first four subjects randomized to treatment arm A.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Group A
Number analyzed (Participants) | 4
h
  Day 1 | 1.75 (0.96)
  Day 14: number analyzed (Participants) | 3
  Day 14 | 1.83 (1.23)

6. Secondary Outcome: Area Under the Concentration-Time Curve [AUC0-6] of CX-4945
Description: To evaluate the area under the concentration-time curve [AUC0-6] of CX-4945 when given at 1000 mg BID PO (Experimental Arm taking CX-4945 only i.e. Group A).
Time Frame: as for outcome 4
Population: Plasma sample of CX-4945 are collected from the first four subjects randomized to treatment arm A.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Group A
Number analyzed (Participants) | 4
h*ng/mL
  Day 1 | 28168.66 (16768.15)
  Day 14: number analyzed (Participants) | 3
  Day 14 | 66147.81 (34540.93)

7. Secondary Outcome: Clinical Benefit of CX-4945 i.e. All-cause Mortality Status - the Number of Deaths Occurred in Each Treatment Group From Randomization (Day 1) Through Day 60
Description: Between the experimental arm with CX-4945 and the control arm, moderate COVID-19 patients' health status will be evaluated in terms of all-cause mortality. Mortality status and cause will be assessed by study staff and the information will be documented on a Clinical Status questionnaire. The data collected will be analyzed at the conclusion of the study to determine if there is a statistically significant difference in all-cause mortality between those whose treatment included CX-4945 and those whose treatment did not include CX-4945.
Time Frame: From Randomization (Day 1) through Day 60
Population: Population: Intent-to-Treat (ITT) Population; The Intent-to-Treat (ITT) population is defined as all randomized subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

8. Secondary Outcome: Clinical Benefit of CX-4945 i.e. Number of Respiratory Failures Occurred in Each Treatment Group From Randomization (Day 1) Through Day 45
Description: Between the experimental arm with CX-4945 and the control arm, moderate COVID-19 patients' health status will be evaluated in terms of the number of respiratory failures. Respiratory failures will be assessed by study staff and the information will be documented on a Clinical Status questionnaire. The information collected will be analyzed at the conclusion of the study to determine if there is a statistically significant difference in number of respiratory failures between those whose treatment included CX-4945 and those whose treatment did not include CX-4945.
Time Frame: From Randomization (Day 1) through Day 45
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

9. Secondary Outcome: Clinical Benefit of CX-4945 i.e. Number of Subjects Hospitalized in Each Treatment Group From Randomization (Day 1) to Day 45
Description: Between the experimental arm with CX-4945 and the control arm, patients will be evaluated in terms of the number of subjects hospitalized in each treatment group. The number of subjects hospitalized will be assessed and the information will be documented on a clinical status questionnaire. The information collected will be analyzed at the conclusion of the study to determine if there is a statistically significant difference in number of subjects hospitalized between those whose treatment included CX-4945 and those whose treatment did not include CX-4945.
Time Frame: From Randomization (Day 1) to Day 45
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
Participants | 1 | 1

10. Secondary Outcome: Clinical Benefit of CX-4945 i.e. Number of Days to Normalization of Oxygen Saturation Level Measured by Pulse Oximeter at Randomization (Day 1), Day 4, Day 8, Day 11, Day 14, Day 28 and Day 45 and Categorized as <96% Versus ≥96%.
Description: Between the experimental arm with CX-4945 and the control arm, patients will be evaluated in terms of time to oxygen saturation level normalization. The information collected will be analyzed at the conclusion of the study to determine if there is a statistically significant difference in time to oxygen saturation level normalization between those whose treatment included CX-4945 and those whose treatment did not include CX-4945. Best Case Scenario = Days to first response for responder, = Days to last observation for non-responder (censored); Worst Case Scenario = Days to first response for responder, = Days to planned last observation date (31 for EQ-5D-5L and SARS-COV-2 Viral Clearance at visit 7, 45 for others at visit 8) for non-responder (censored); Days to first response = date of first response - the first treatment date/time + 1 Days to last observation = date of last evaluation - the first treatment date/time + 1 For Arm SOC, the first treatment date is the date of visit 2.
Time Frame: Randomization (Day 1), Day 4, Day 8, Day 11, Day 14, Day 28 and Day 45
Population: as for outcome 7
Measure: Mean (Standard Error); unit: days
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
days
  Best Case Scenario: number analyzed (Participants) | 9 | 10
  Best Case Scenario | 2 (0.7) | 4 (1.4)
  Worst Case Scenario: number analyzed (Participants) | 9 | 10
  Worst Case Scenario | 2 (0.7) | 4 (1.4)

11. Secondary Outcome: Clinical Benefit of CX-4945 i.e. Proportion of Subjects With Disease Progression or Improvement in Health Status Occurring From Randomization (Day 1) to Day 28.
Description: Between the experimental arm with CX-4945 and the control arm, proportion of subjects with disease progression or improvement in health status occurring from Randomization (Day 1) to Day 28 will be evaluated. Disease progression is defined as change in subject health status assessment from item 7 to items 1- 6 and health improvement -as change from item 7 to item 8, evaluated by the ordinal NIAID 8- point Clinical Progression Outcomes scale - collected at every visit from randomization (Day 1) through Day 45. The information collected will be analyzed at the conclusion of the study to determine if there is a statistically significant difference in clinical status between those whose treatment included CX-4945 and those whose treatment did not include CX-4945.
Time Frame: From Randomization (Day 1) to Day 28
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
Participants
  Baseline to Visit 7 (Day 28): number analyzed (Participants) | 8 | 10
  Baseline to Visit 7 (Day 28): Improvement | 6 | 7
  Baseline to Visit 7 (Day 28): Progression | 0 | 0
  Baseline to Visit 7 (Day 28): Else | 2 | 3
  Baseline to Visit 8 (Day 45), LOCF: number analyzed (Participants) | 8 | 10
  Baseline to Visit 8 (Day 45), LOCF: Improvement | 6 | 6
  Baseline to Visit 8 (Day 45), LOCF: Progression | 0 | 0
  Baseline to Visit 8 (Day 45), LOCF: Else | 2 | 4

12. Secondary Outcome: Clinical Benefit of CX-4945 i.e. Changes in the Total Score for Q1~Q5 of the EQ-D5-5L From Randomization (Day 1) to Day 8, Day 14 and Day 28.
Description: Changes in the total score for Q1~Q5 of the EQ-D5-5L (used as an indicator of symptom improvement) from Baseline (Day 1) to Day 8, 14, 28 were evaluated. The 5-level EQ-5D version (EQ-5D-5L) was used to assess five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Four times during the study (baseline, Day 8, Day 14 and Day 28) the patients were asked to complete health status survey by answering 6 questions about their health and quality of life. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Patients were also asked to assess their overall health status by selecting a number between 1 and 100 to describe the condition of their health, 100 being the best imaginable.
Time Frame: From randomization (Day 1) to Day 8, Day 14 and Day 28.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
score on a scale
  Visit 4 (Day 8) - Visit 2 (Day 1) | -2.2 (2.39) | -1.3 (2.67)
  Visit 6 (Day 14, EOT) - Visit 2 (Day 1): number analyzed (Participants) | 10 | 9
  Visit 6 (Day 14, EOT) - Visit 2 (Day 1) | -3.0 (2.31) | -3.3 (2.00)
  Visit 7 (Day 28, F1), LOCF - Visit 2 (Day 1): number analyzed (Participants) | 8 | 10
  Visit 7 (Day 28, F1), LOCF - Visit 2 (Day 1) | -3.5 (0.93) | -3.9 (2.88)

13. Secondary Outcome: Clinical Benefit of CX-4945 i.e. Changes in the Imaginable Health Status of the EQ-D5-5L From Randomization (Day 1) to Day 8, Day 14 and Day 28.
Description: Changes in the Imaginable Health Status of the EQ-D5-5L (used as an indicator of symptom improvement) from Baseline (Day 1) to Day 8, 14, 28 were evaluated. The 5-level EQ-5D version (EQ-5D-5L) was used to assess five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Four times during the study (baseline, Day 8, Day 14 and Day 28) the patients were asked to complete health status survey by answering 6 questions about their health and quality of life. Patients were also asked to assess their overall health status by selecting a number between 1 and 100 to describe the condition of their health, 100 being the best imaginable.
Time Frame: From randomization (Day 1) to Day 8, Day 14 and Day 28.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
score on a scale
  Visit 4 (Day 8) - Visit 2 (Day 1) | 15.7 (11.80) | 16.5 (7.09)
  Visit 6 (Day 14, EOT) - Visit 2 (Day 1) | 24.1 (12.40) | 30.3 (11.87)
  Visit 7 (Day 28, F1), LOCF - Visit 2 (Day 1): number analyzed (Participants) | 8 | 10
  Visit 7 (Day 28, F1), LOCF - Visit 2 (Day 1) | 28.8 (19.83) | 39.5 (9.85)

14. Secondary Outcome: CX-4945 Inflammatory Marker Outcomes i.e. Plasma IL-6
Description: Labs to evaluate changes in plasma IL-6 (interleukin-6 in ng/L) levels between the patients within the experimental arm with CX-4945 and the control arm, of patients with moderate COVID-19. The information collected will be analyzed at the conclusion of the study to determine if there is a statistically significant difference in plasma IL-6 levels between those whose treatment included CX-4945 and those whose treatment did not include CX-4945.
Time Frame: Changes in plasma IL-6 level from Randomization (Day 1) to Day 4, Day 8, Day 11, and Day 14.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
ng/L
  Adjusted Visit 3 (Day 4) - Baseline: number analyzed (Participants) | 4 | 4
  Adjusted Visit 3 (Day 4) - Baseline | 1.43 (1.511) | -2.73 (6.784)
  Adjusted Visit 4 (Day 8) - Baseline: number analyzed (Participants) | 3 | 3
  Adjusted Visit 4 (Day 8) - Baseline | 25.08 (39.828) | 2.83 (5.550)
  Adjusted Visit 5 (Day 11) - Baseline: number analyzed (Participants) | 3 | 2
  Adjusted Visit 5 (Day 11) - Baseline | -14.35 (27.882) | 0.40 (4.363)
  Adjusted Visit 6 (Day 14) - Baseline: number analyzed (Participants) | 3 | 1
  Adjusted Visit 6 (Day 14) - Baseline | -23.47 (34.018) | -10.06 (NA) — In the CSR, 'M' is noted in the SD column likely indicates extensive missing data, with 1 analyzed and 9 missing.

15. Secondary Outcome: CX-4945 Inflammatory Marker Outcomes i.e. Plasma CRP
Description: Labs to evaluate changes in plasma CRP (C-reactive protein in mg/DL) levels between the patients within the experimental arm with CX-4945 and the control arm, of patients with moderate COVID-19. The information collected will be analyzed at the conclusion of the study to determine if there is a statistically significant difference in plasma CRP levels between those whose treatment included CX-4945 and those whose treatment did not include CX-4945.
Time Frame: Changes in CRP from randomization (Day 1) to Day 4, Day 8, Day 11, and Day 14.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
mg/dL
  Adjusted Visit 3 (Day 4) - Baseline: number analyzed (Participants) | 6 | 6
  Adjusted Visit 3 (Day 4) - Baseline | 0.17 (0.261) | -0.40 (1.752)
  Adjusted Visit 4 (Day 8) - Baseline: number analyzed (Participants) | 5 | 6
  Adjusted Visit 4 (Day 8) - Baseline | -0.14 (0.622) | -0.61 (1.508)
  Adjusted Visit 5 (Day 11) - Baseline: number analyzed (Participants) | 5 | 6
  Adjusted Visit 5 (Day 11) - Baseline | -0.77 (1.513) | -0.59 (1.379)
  Adjusted Visit 6 (Day 14) - Baseline: number analyzed (Participants) | 6 | 6
  Adjusted Visit 6 (Day 14) - Baseline | -0.72 (1.597) | -0.51 (1.520)

16. Secondary Outcome: CX-4945 Inflammatory Marker Outcomes i.e. Plasma LDH
Description: Labs to evaluate changes in plasma LDH (lactic acid dehydrogenase in U/L) levels between the patients within the experimental arm with CX-4945 and the control arm, of patients with moderate COVID-19. The information collected will be analyzed at the conclusion of the study to determine if there is a statistically significant difference in plasma LDH levels between those whose treatment included CX-4945 and those whose treatment did not include CX-4945.
Time Frame: Changes in LDH from randomization (Day 1) to Day 4, Day 8, Day 11, and Day 14.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
U/L
  Adjusted Visit 3 (Day 4) - Baseline: number analyzed (Participants) | 9 | 7
  Adjusted Visit 3 (Day 4) - Baseline | 7.11 (23.661) | 48.71 (97.324)
  Adjusted Visit 4 (Day 8) - Baseline: number analyzed (Participants) | 9 | 7
  Adjusted Visit 4 (Day 8) - Baseline | 28.78 (122.942) | 47.57 (100.565)
  Adjusted Visit 5 (Day 11) - Baseline: number analyzed (Participants) | 6 | 7
  Adjusted Visit 5 (Day 11) - Baseline | -29.17 (79.200) | 12.86 (34.868)
  Adjusted Visit 6 (Day 14) - Baseline: number analyzed (Participants) | 9 | 6
  Adjusted Visit 6 (Day 14) - Baseline | -6.67 (98.659) | 50.00 (87.088)

17. Secondary Outcome: CX-4945 Inflammatory Marker Outcomes i.e. Plasma CPK
Description: Labs to evaluate changes in plasma CPK (creatine phosphokinase in U/L) levels between the patients within the experimental arm with CX-4945 and the control arm, of patients with moderate COVID-19. The information collected will be analyzed at the conclusion of the study to determine if there is a statistically significant difference in plasma CPK levels between those whose treatment included CX-4945 and those whose treatment did not include CX-4945.
Time Frame: Changes in CPK from randomization (Day 1) to Day 4, Day 8, Day 11, and Day 14.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
U/L
  Adjusted Visit 3 (Day 4) - Baseline: number analyzed (Participants) | 9 | 8
  Adjusted Visit 3 (Day 4) - Baseline | 6.11 (64.297) | -14.50 (36.154)
  Adjusted Visit 4 (Day 8) - Baseline: number analyzed (Participants) | 9 | 8
  Adjusted Visit 4 (Day 8) - Baseline | 11.89 (116.393) | -12.13 (24.908)
  Adjusted Visit 5 (Day 11) - Baseline: number analyzed (Participants) | 7 | 8
  Adjusted Visit 5 (Day 11) - Baseline | -30.14 (72.073) | -17.25 (25.811)
  Adjusted Visit 6 (Day 14) - Baseline: number analyzed (Participants) | 9 | 7
  Adjusted Visit 6 (Day 14) - Baseline | -23.56 (64.211) | -16.86 (31.882)

18. Secondary Outcome: CX-4945 Inflammatory Marker Outcomes i.e. Plasma Ferritin
Description: Labs to evaluate changes in plasma ferritin (μg/L) levels between the patients within the experimental arm with CX-4945 and the control arm, of patients with moderate COVID-19. The information collected will be analyzed at the conclusion of the study to determine if there is a statistically significant difference in plasma ferritin levels between those whose treatment included CX-4945 and those whose treatment did not include CX-4945.
Time Frame: Changes in ferritin from randomization (Day 1) to Day 4, Day 8, Day 11, and Day 14.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
μg/L
  Adjusted Visit 3 (Day 4) - Baseline: number analyzed (Participants) | 8 | 6
  Adjusted Visit 3 (Day 4) - Baseline | -18.35 (44.322) | 2.02 (5.454)
  Adjusted Visit 4 (Day 8) - Baseline: number analyzed (Participants) | 9 | 7
  Adjusted Visit 4 (Day 8) - Baseline | -57.52 (175.573) | -37.99 (73.496)
  Adjusted Visit 5 (Day 11) - Baseline: number analyzed (Participants) | 7 | 7
  Adjusted Visit 5 (Day 11) - Baseline | -90.07 (251.589) | -63.03 (76.342)
  Adjusted Visit 6 (Day 14) - Baseline: number analyzed (Participants) | 9 | 7
  Adjusted Visit 6 (Day 14) - Baseline | -152.12 (421.528) | -79.10 (96.784)

19. Secondary Outcome: CX-4945 Inflammatory Marker Outcomes i.e. Plasma D-Dimer
Description: Labs to evaluate changes in plasma D-dimer (μg/mL) levels between the patients within the experimental arm with CX-4945 and the control arm, of patients with moderate COVID-19. The information collected will be analyzed at the conclusion of the study to determine if there is a statistically significant difference in plasma D-dimer levels between those whose treatment included CX-4945 and those whose treatment did not include CX-4945.
Time Frame: Changes in D-dimer from randomization (Day 1) to Day 4, Day 8, Day 11, and Day 14.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
μg/mL
  Adjusted Visit 3 (Day 4) - Baseline: number analyzed (Participants) | 6 | 6
  Adjusted Visit 3 (Day 4) - Baseline | 0.00 (0.118) | -0.21 (0.544)
  Adjusted Visit 4 (Day 8) - Baseline: number analyzed (Participants) | 3 | 5
  Adjusted Visit 4 (Day 8) - Baseline | -0.10 (0.164) | 0.13 (0.152)
  Adjusted Visit 5 (Day 11) - Baseline: number analyzed (Participants) | 4 | 2
  Adjusted Visit 5 (Day 11) - Baseline | -0.08 (0.138) | -0.01 (0.007)
  Adjusted Visit 6 (Day 14) - Baseline: number analyzed (Participants) | 1 | 4
  Adjusted Visit 6 (Day 14) - Baseline | -0.04 (NA) — In the CSR, 'M' is noted in the SD column likely indicates extensive missing data, with 1 analyzed and 9 missing. | -0.09 (0.170)

ADVERSE EVENTS:
Time Frame: From randomization (Day 1) to Day 60
Description: Adverse events occurring from randomization (Day 1) to Day 60 (including vital signs, physical findings, clinical laboratory, and ECG results) as characterized by type, frequency, severity [(as graded by Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (https://www.fda.gov/media/73679/download)], timing, seriousness, and relationship to study therapy.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/10
Other Adverse Events (participants affected / at risk) | 8/10 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=10) | Group B (N=10)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=10) | Group B (N=10)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dyschezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis viral (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1)
Glucose urine present (Investigations) | 1 (1) | 0 (0)
Haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0)
Urine analysis abnormal (Investigations) | 2 (2) | 0 (0)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT04663737/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT04663737/SAP_001.pdf